CLINICAL TRIAL: NCT00609037
Title: A Pilot/Feasibility Study on Wound Repair and Body Contouring Surgery After Gastric By-pass
Brief Title: Wound Repair and Body Contouring Surgery After Gastric Bypass
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kevin Hagan, Associate Professor, Vanderbilt University
Other Study IDs: 050298
Record Dates: First submitted 2008-01-25; First posted 2008-02-06 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Obesity, Morbid
Keywords: Gastric Bypass; Body contouring; Excessive weight loss
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Individuals who has had a weight reduction procedure such as gastric bypass and have body contouring surgery to remove the excessive skin due to the weight loss
- 2: Normal controls include individuals who schecule to have an abdominoplasty and are within normal for height and weight

SUMMARY:
The primary aim of our study is to test the hypothesis that wound healing is impaired in the patient who has experienced massive weight reduction following gastric bypass for morbid obesity. Specifically we will document post-surgical local complications and evaluate multiple wound healing parameters in two patient populations in a prospective fashion. The test group will consist of patients who have undergone dramatic weight loss and are much in need of a panniculectomy due to excessive skin redundancy. The control group will consist of patients within normal weight ranges who are seeking an abdominoplasty.

DETAILED DESCRIPTION:
The morbidly obese patient after successful weight reduction surgery represents a poorly understood patient population that presents unique quandaries. Prior to gastric bypass surgery, many of these patients have Type II diabetes, frequent skin infections from poor hygiene, and multiple medical co-morbidities. Fortunately, numerous problems resolve during the period of the rapid weight loss. Typically the Type II diabetes comes under control without medication and patients experience improvement in mobility and psychosocial adjustment. Unfortunately new dilemmas can rise such as vitamin deficiencies due to many months of starvation, residual end glycosylation products in diabetic skin and massive skin redundancies in multiple locations. Excessive skin is prone to infection. Patients continue to be plagued with postural problems, functional problems (improper personal hygiene, continued difficulties in ambulation) and psychosocial problems associated with a poor body image. Body contouring can provide such patients with marked improvements in lifestyle. The post-bariatric patient population is rapidly increasing in number, yet their wound healing responses to accidental or surgical trauma are unreported in the literature.

Recent studies have documented clinical suspicions that the post-bariatric patient is at an increased risk for wound healing complications following body contouring procedures. The most recent retrospective study of 30 patients

assessed post-surgical outcomes following body contouring procedures in multiple body locations and noted a 20% incidence of wound breakdown and a 16% incidence of seroma (1). An earlier retrospective study comparing panniculectomy in post bariatric patients to those receiving a simultaneous panniculectomy plus gastric bypass documented wound infections (16%), dehiscence (13%) and skin necrosis (6%) in the post bariatric group (2). A prospective study of ten post-bariatric patients who were given a circumferential abdominoplasty likewise experienced wound complications: (33% seromas, 16.6% dehiscence, and infections 8.2%) (3). An 11 patient dermalipectomy series for body contouring after bariatric surgery showed a 27% incidence of infection and seroma (4). To date, the highest rate of wound healing complications was reported in 46 out of 55 (86%) dermolipectomy patients (5). Taken together these reports provide clinical evidence that wound healing is impaired in the post-bariatric patient population. We are prepared to undertake a quantitative evaluation of wound repair characteristics in this select population.

There are multiple reasons to suspect that the skin itself may be defective in these patients who have undergone massive weight reduction. A lifetime of stretched out skin can thin the density of epidermal appendages and peripheral nerve endings, alter the vascular network, diminish the elasticity and alter the weave of the collagen bundles in the reticular dermis. Such negative circumstances may impede the delivery of oxygen and nutrients and ultimately hinder tensile strength. Nutritional deficiencies from the forced starvation are thought to decrease anabolic processes and impair the inflammatory processes, factors that also govern the timing and quality of wound repair. Dehiscence rates could be negatively impacted by this synergy of alterations. While the post-bariatric patients can electively seek body contouring surgery, it is certain that the ever increasing number of post-bariatric patients will experience unexpected trauma or non-elective surgical procedures - all circumstances that also challenge the body to repair itself. We maintain that it will be important to document wound healing deficiencies so that optimal treatment plans can be implemented when the need arises.

Disclaimer: Individuals who participate in this study are financially responsible for all costs relating to the surgery!

ELIGIBILITY:
Inclusion Criteria:

* Gastric Bypass or other weight reduction procedure requesting body contouring surgery
* Cosmetic abdominoplasty
* Be willing to complete study required bloodwork and collection of tissue and fluid samples

Exclusion Criteria:

* Unable to comply with study requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All potential subjects presenting to the plastic surgery practice ages 18-65 will be approached for participation
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2006-01; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Number and type of wound healing complications in the panniculectomy group compared to the control group | 1,5,14, 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Marcia E Spear, MSN, Study Director — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States